CLINICAL TRIAL: NCT06677385
Title: Effect of Low-Level Laser on Crevicular Interleukin-1β Concentration in Patients With Periodontal Disease: A Relation to Periodontal Inflammaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Asmaa EssamEldin Ahmed, Teaching assistant, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022/0082
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-11

CONDITIONS: Periodontal Diseases; Old Age
MeSH Terms: conditions — Periodontal Diseases | interventions — Lasers, Semiconductor; Debridement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Conventional scaling and debridement in young aged patients (Experimental): scaling and debridement
  Interventions: Procedure: conventional scaling and debridement
- Conventional scaling and debridement of old aged patients (Experimental)
  Interventions: Procedure: conventional scaling and debridement
- diode laser as adjunctive to conventional scaling and debridement for old age patients (Experimental)
  Interventions: Radiation: diode laser as adjunctive to conventional scaling and debridement
- diode laser as adjunctive to conventional scaling and debridement for young age patients (Experimental)
  Interventions: Radiation: diode laser as adjunctive to conventional scaling and debridement

INTERVENTIONS:
Radiation: diode laser as adjunctive to conventional scaling and debridement — diode laser as adjunctive to conventional scaling and debridement for old age patients
  Arms: diode laser as adjunctive to conventional scaling and debridement for old age patients; diode laser as adjunctive to conventional scaling and debridement for young age patients
Procedure: conventional scaling and debridement — conventional scaling and debridement
  Arms: Conventional scaling and debridement in young aged patients; Conventional scaling and debridement of old aged patients

SUMMARY:
This study is done to compare between young age and old age patients with periodontitis (inflammaging) and the effect of diode laser as adjunctive to scaling and debridement

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Aged below 40 or above 60.
3. Provide informed consent and willingness to cooperate with study protocol.
4. Periodontitis stage II patients:

   * CAL from 3-4 mm.
   * Radiographic bone loss (15% to 33%).
   * No tooth loss due to periodontitis.
   * Maximum probing depth ≤ 5 mm, mostly horizontal bone loss

Exclusion Criteria:

1. Patients with heavy smoking habits
2. History of antibiotics in the previous three months.
3. Pregnant or lactating female.
4. Treatment with any systemic drug.
5. History of systemic disease.
6. Patients who received periodontal treatment in the last 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Gingival index | first visit, second follow up after 1 month and final follow up after 6 months
Clinical attachment loss | first visit, second follow up after 1 month and final follow up after 6 months
Interleukin 1 beta | first visit, second follow up after 1 month and final follow up after 6 months
  collected and analyzed by ELISA from Gingival crevicular fluid and blood serum

CONTACTS AND LOCATIONS:
Locations (1):
- Misr University foe Science and Technology, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided